CLINICAL TRIAL: NCT04741282
Title: Effect of Pulmonary Tele-rehabilitation With and Without Progressive Muscle Relaxation Program in Covid-19 Patients After Hospital Discharge: Randomized Clinical Trial
Brief Title: Pulmonary Tele-rehabilitation and Progressive Muscle Relaxation on Discharged Covid-19 Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 18225
Record Dates: First submitted 2021-01-30; First posted 2021-02-05 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pulmonary telerehabilitation plus progressive muscle relaxation training (Experimental): This group will perform six week pulmonary rehabilitation program and progressive muscle relaxation exercise at theirs home, with two supervised sessions by physiotherapist per week via videoconferencing.
  Interventions: Other: Pulmonary telerehabilitation; Other: progressive muscle relaxation training
- pulmonary telerehabilitation (Active Comparator): This group will perform six week pulmonary rehabilitation program at theirs home, with two supervised sessions by physiotherapist per week via videoconferencing.
  Interventions: Other: Pulmonary telerehabilitation

INTERVENTIONS:
Other: Pulmonary telerehabilitation — pulmonary telerehabilitation program include breathing exercise,aerobics exercise and upper and lower limbs muscle strengthening exercise
Other: progressive muscle relaxation training — summarized Jacobson progressive muscle relaxation training method
  Arms: pulmonary telerehabilitation plus progressive muscle relaxation training

SUMMARY:
The aim of this study is to investigate efficacy of internet based pulmonary rehabilitation and progressive muscle relaxation program on functional capacity, depression and anxiety, dyspnea, fatigue, sleep quality and quality of life in covid19 patients after hospital discharge

DETAILED DESCRIPTION:
Novel coronavirus disease 2019 (covid19) could cause respiratory and physical dysfunction, anxiety and depression, fatigue and affect sleep quality and quality of life in infected patient after hospital discharge. there is expect that pulmonary rehabilitation can improve these symptoms and prevent complications in these cases. It seems that Progressive muscle relaxation exercise could improve pulmonary rehabilitation effect. Due to social isolation of Covid 19 patients after hospital discharge, internet base rehabilitation will be used in this study. participants will be randomized in two pulmonary tele-rehabilitation groups after hospital discharge. One group will be received pulmonary rehabilitation include education, breathing exercises, aerobic and upper and lower limbs muscle strengthening exercises. Another group will be perform progressive muscle relaxation in addition of these exercise. Treatment duration is 6 week with 5 days/week frequency. Two exercise sessions per week will be supervised with expert physiotherapist via videoconferencing.

Outcomes will be measured at baseline, within two week and at the end of six week exercises program.

ELIGIBILITY:
Inclusion Criteria:

* Covid 19 patient that confirmed with polymerase chain reaction test (PCR)
* Hospitalized Corvid 19 patients after discharge
* Accessibility to internet and using video call

Exclusion Criteria:

* Mental and physical disability
* Uncontrolled cardiac dysfunction such as arrhythmia
* Sever neurological condition such as guillain-barre and stroke
* Uncontrolled diabetes or blood pressure
* Pregnant women
* Re-hospitalization during treatment program
* Chronic pulmonary and kidney condition

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Functional capacity | change from baseline in 6MWT at 2 and 6 weeks
  six minute walk test (6MWT)

SECONDARY OUTCOMES:
dyspnea | change from baseline in Borg scale at 2 and 6 weeks
  Borg scale, The borg scale is a self-rating tool to measure the degree of breathlessness on a scale from 0 to 10, higher score mean worse dyspnea
Sleep quality | change from baseline in PSQI at 6 week
  petersburg sleep quality index (PSQI), PSQI is a eighteen item scale.The total scores range is 0-21. A higher score indicates a worse sleep quality.
anxiety and depression | change from baseline in HADS at 6 week
  hospital anxiety and depression scale (HADS), HADS is a fourteen item scale. Seven of the items relate to anxiety and seven relate to depression.The total scores range is 0-21 for both depression and anxiety scores. A higher score indicates a worse depression and anxiety.

OTHER OUTCOMES:
health status | change from baseline in SGRQ at 6 week
  St. George's Respiratory Questionnaire (SGRQ), Three component scores are calculated for the SGRQ (symptom,activity, impact). Scores are expressed as a percentage of overall impairment where 100 represents worst possible health status and 0 indicates best possible health status.
fatigue | change from baseline in FSS at 2 and 6 weeks
  fatigue severity scale (FSS). FSS is nine item scale. the total score range is 1-7. a higher score indicates a worse fatigue severity.
Quality of life and well-being | change from baseline in SF36 at 6 week
  Quality of life will measure using SF-36 questionnaire, SF-36 is a 36 item scale.The total scores range is 0-100. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Javad Sarrafzadeh, PhD, Study Chair — Department of Physiotherapy, School of Rehabilitation Sciences, Iran University of Medical Sciences
Locations (1):
- Iran university of medical sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No